CLINICAL TRIAL: NCT07036770
Title: Coronary Evaluation And Guided Lesion Exploration Using Photon-counting CT and Intracoronary Imaging Techniques
Acronym: C-EAGLE
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S70500
Record Dates: First submitted 2025-05-26; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease; OCT Angiography; CT
Keywords: PCCT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coronary CT scan using photon-counting CT — A dedicated cardiac UHR PCCT will be conducted within a maximum of 24 hours in ACS subjects and 72 hours in CCS subjects prior to the invasive CAG. Additionally, patients are also eligible for inclusion in case no PCCT is conducted prior to CAG, as long as no PCI is performed during the initial CAG. In these cases, the PCCT must be conducted within 24 hours for ACS patients and within 72 hours for CCS patients.

SUMMARY:
This study evaluates the diagnostic accuracy and limitations of photon-counting computed tomography (PCCT) in characterizing coronary plaque, with comparisons to optical coherence tomography (OCT) and intravascular ultrasound (IVUS). The objective is to assess whether cardiac ultra-high resolution (UHR) PCCT -with its improved spatial resolution and superior soft tissue contrast relative to conventional CT- can serve as a reliable, non-invasive alternative for coronary plaque assessment and support clinical decision-making. A total of 100 patients with either acute or chronic coronary syndrome will be enrolled, including 40 individuals with suspected in-stent restenosis and 10 patients one year post-percutaneous coronary intervention (PCI) for chronic total occlusion (CTO). All participants will undergo invasive coronary angiography based on current European Society of Cardiology guidelines. Cardiac PCCT imaging will be conducted shortly before the angiographic procedure, accompanied by invasive OCT evaluation. Additionally, a subgroup of 10 patients will undergo both OCT and IVUS, allowing for direct comparison across imaging modalities. OCT, regarded as the gold standard for plaque characterization, offers near-histological resolution for identifying plaque features, while IVUS is particularly effective in evaluating plaque burden and volume.

ELIGIBILITY:
Inclusion criteria:

Participants eligible for inclusion in this study must meet all of the following criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures.
2. At least 18 years of age at the time of signing the Informed Consent Form (ICF).
3. Patients presenting with suspected acute coronary syndrome (UA or NSTEMI) or chronic coronary syndrome (stable angina or silent ischemia).

Exclusion criteria:

Participants eligible for this study must not meet any of the following criteria:

1. Patients presenting with STEMI.
2. Haemodynamically unstable patients.
3. Unstable ventricular arrhythmias.
4. Killip class III-IV heart failure.
5. Creatinine clearance <30 ml/min/1.73 m2 (as calculated by CKD-EPI formula 2009 for estimated GFR) and not on dialysis. Note: patients dependent on long-term dialysis are eligible for enrolment irrespective of their creatinine clearance levels.
6. Severe coronary vessel tortuosity.
7. Subject has known hypersensitivity to radiocontrast dye or that cannot be adequately pre-medicated.
8. Female who is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to enrol 100 patients with acute or chronic coronary syndrome, including 40 participants with suspected in-stent restenosis and 10 participants one year after a CTO PCI.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of coronary PCCT angiography. | From PCCT until OCT run, completed within 72 hours.
  Assessment of co-primary endpoints luminal area (mm²), stenosis grade (%) and plaque content (mm²) of coronary PCCT as compared to OCT imaging.

SECONDARY OUTCOMES:
High-risk plaque features. | From PCCT until OCT run, completed within 72 hours.
  Correlation of high-risk features on coronary PCCT with OCT findings, including presence of TCFA, lipid-rich plaque, macrophages, spotty calcification, microvessels, cholesterol crystal and/or layered plaque.
Plaque volume. | From PCCT until IVUS run, completed within 72 hours.
  Comparison between plaque volume on coronary PCCT and IVUS (mm³).
Coronary reconstruction algorithm. | From PCCT until OCT run, completed within 72 hours.
  Analysis of coronary artery reconstruction algorithm with PCCT as compared to invasive coronary angiogram (minimal lumen area; mm²).

CONTACTS AND LOCATIONS:
Overall Officials: Tom Adriaenssens, MD PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided